CLINICAL TRIAL: NCT01650883
Title: A Randomized Prospective Open-label Comparison of Two Vitamin D3 Repletion Strategies in Vitamin D Deficient Patients
Brief Title: A Prospective Open-label Comparison of Two Vitamin D3 Repletion Strategies in Vitamin D Deficient Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VitD3USFstudy
Record Dates: First submitted 2012-07-23; First posted 2012-07-26 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: Vitamin D 25 OH Deficiency
Keywords: Vitamin D3; Vitamin D 25 OH
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cholecaliferol 50,000 IU PO Q10 days x 40 days (Experimental): Patients in this arm receive Cholecalciferol (vitamin D3) via PO route every 10 days for 40 days for a total of 200,000 IU of Vitamin D3. They also receive daily 1200 mg of Calcium Carbonate via PO route daily for 40 days.
  Interventions: Dietary Supplement: Cholecalciferol
- Cholecalciferol 5,000 IU PO daily x 40 days (Experimental): Patients in this arm receive 5,000 IU of Cholecalciferol (Vitamin D3) via PO route daily for 40 days for a total of 200,000 IU. These patients also receive 1200 mg of daily Calcium Carbonate via PO route for 40 days.
  Interventions: Dietary Supplement: Cholecalciferol 5,000 IU

INTERVENTIONS:
Dietary Supplement: Cholecalciferol — Cholecalciferol 50,000 IU PO every 10 days for 40 days
  Other Names: Vitamin D3
  Arms: Cholecaliferol 50,000 IU PO Q10 days x 40 days
Dietary Supplement: Cholecalciferol 5,000 IU — Cholecalciferol 5,000 IU PO daily for 40 days + 1200 mg Calcium Carbonate PO daily for 40 days.
  Other Names: Vitamin D3
  Arms: Cholecalciferol 5,000 IU PO daily x 40 days

SUMMARY:
The purpose of this study is to determine whether one of two Vitamin D3 (cholecalciferol) oral treatment regimens is superior to the other in normalizing Vitamin 25 OHD serum levels. While these two regimens in the end provide equal total dosing, the two arms differ in frequency and dosing during a 40 day treatment plan. The primary endpoint will be a direct comparison of two dosing regimens of Vitamin D3 repletion at day 40 (+/- 3 days) using a paired T-test. Secondary endpoints include record of adverse events throughout the 40 day study period as well as changes in basic laboratory values including CMP and ionized Calcium.

The investigators hypothesize that the Cholecalciferol (Vitamin D3) daily dosing arm of 5000 IU daily will result in more efficient replacement as compared to the 50,000 IU dosing given every 10 days. Our goal will be to achieve a serum Vitamin 25 OH D level of > 50 mg/dL at day 40. The investigators propose that 75% of the subjects on daily Vitamin D3 will achieve this level and that 35% of the subjects in the every 10 days dosing arm will reach this goal.

DETAILED DESCRIPTION:
This is a 40 day randomized prospective open-label study of two arms of vitamin D repletion protocols. USF clinic patients seen in the Rheumatology clinic, who meet criteria and have a baseline vitamin 25 OH D level of less than or equal to 32 mg/dL, will be randomized to two treatment arms. A Vitamin 25 OH D level of less than 32 mg/dL but above 20 mg/dL will be defined as insufficient. Similarly, a vitamin 25 OH D level of less than or equal to 20 mg/dL will be defined as deficient.

Patients in arm one will be repleted with Cholecalciferol (Vitamin D3) at 5000 IU orally daily for 40 days. Arm two of this treatment protocol will consist of 50,000 IU cholecalciferol (Vitamin D3) orally every 10 days starting on day 1 for 40 days. All subjects in both groups will receive a total dose of 200,000 IU of Vitamin D3 after 40 days of treatment. Each patient will also receive oral supplementation of 1200 mg daily calcium carbonate. Patients will return to clinic on day 40 (+/- 3 days) for a follow up serum vitamin 25 OH D and Calcium level. Compliance will be checked at that time with a pill count.

Clinical Significance: This trial asks the question as to whether one oral repletion therapy is superior to another in a 40 day time period. Given that current standard of care is based on individual practitioner experience, it may be beneficial for a standard protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - open ended to both males and females
* Able to give informed consent
* 25 OH-Vitamin D level of < or = 32 mg/dL
* Creatinine of < 1.9 or Creatinine Clearance (CrCl) of greater than or equal to 40 mL/min/1.73 m^2.
* English speaking

Exclusion Criteria:

* Creatinine of greater to or equal to 1.9 or CrCl less than 40 mL/min/1.73 m^2 (as calculated on MDRD.com)
* History of hyperparathyroidism, a known risk factor for hyperkalemia
* History of nephrolithiasis given that hypervitaminosis D can increase the risk of nephrolithiasis
* Current use of any dose of glucocorticoids, a known risk factor for hypercalcuria
* History of sarcoidosis, tuberculosis, or Paget's disease which are known risk factors for hypercalcemia
* (Random) Molar Calcium:Creatinine urinary concentration of > 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2009-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be a direct comparison of two dosing regimens of Vitamin D3 repletion at day 40 (+/- 3 days) using a paired sample T-test by measuring the change in Vitamin D 25 OH from baseline to day 40 of treatment for both treatment groups. | 40 days +/- 3 days

SECONDARY OUTCOMES:
Adverse events throughout the 40 day study | 40 +/- 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Julio Gonzalez, MD, Principal Investigator — University of South Florida College of Medicine; John D Carter, MD, Principal Investigator — University of South Florida Division of Rheumatology
Locations (1):
- University of South Florida, Tampa, Florida, United States